CLINICAL TRIAL: NCT02086864
Title: A Randomized, Double Blind, Placebo Controlled Study of Homeopathic Treatment of Children and Youth With Attention Deficit Hyperactivity Disorder
Brief Title: A Placebo Controlled Study of Homeopathic Treatment of Children and Youth With ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Lotte & John Hecht Memorial Foundation (Other); Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Heather Boon, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UToronto-29722; 079-2013 (Other: Centre for Addiction and Mental Health)
Record Dates: First submitted 2014-03-07; First posted 2014-03-13 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; Homeopathy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lactose; Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual care (No Intervention)
- Individualized homeopathic medicine treatment (Active Comparator): Participant will have a homeopathic consultation and be given a homeopathic medicine. Homeopathic medicines are chosen from those available for sale in Canada.
  Interventions: Drug: lactose/sucrose granule (Individualized homeopathic medicine treatment); Behavioral: Homeopathic consultation
- Unmedicated lactose/sucrose pill (Placebo Comparator): Participant will receive a homeopathic consultation and receive an unmedicated lactose/sucrose pill.
  Interventions: Drug: Placebo lactose/sucrose pill; Behavioral: Homeopathic consultation

INTERVENTIONS:
Drug: lactose/sucrose granule (Individualized homeopathic medicine treatment) — The homeopathic remedy (study medication) for each patient will be chosen from among the homeopathic medicines manufactured by Boiron Canada and currently approved for sale in Canada by Health Canada. As per classical homeopathy practice, once the most appropriate homeopathic remedy has been chosen, it will be prescribed by the homeopath according to her/his clinical judgment (maximum on a daily basis, 3 times per day, minimum 1 dose (or zero doses on the second consult or later)) with administration instructions given to the parent and patient as appropriate. Water dosing, in which a lactose/sucrose granule remedy is dissolved in 250 ml of water will be used based on the homeopath's clinical judgment. Only one remedy will be administered at a time.
  Arms: Individualized homeopathic medicine treatment
Drug: Placebo lactose/sucrose pill
  Arms: Unmedicated lactose/sucrose pill
Behavioral: Homeopathic consultation
  Other Names: Homeopathic case taking (90 minutes)
  Arms: Individualized homeopathic medicine treatment; Unmedicated lactose/sucrose pill

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is a developmental disorder that presents during childhood, with at least some symptoms causing impairment before the age of seven. It is characterized by developmentally inappropriate levels of inattention and/or hyperactive-impulsive behavior, with significant impairment occurring in at least two settings. It affects approximately 5.2 million children in the United States. Homeopathic treatment has been shown to be a promising intervention for ADHD, however the reasons for that effectiveness is unclear. Specifically, it is unclear whether improvement is due to the homeopathic medicine, the consultative process, or other non-specific effects.

This study has 3 primary objectives: 1. to determine if there are any specific effects of homeopathic medicines in the treatment of ADHD, 2. to determine if there any specific effects the homeopathic consultation alone in the treatment of ADHD, and 3. to determine if there is an overall effect of homeopathic treatment (homeopathic medicines plus consultation) in the treatment of ADHD.

This is a three arm study. Participants will be randomized to one of three arms:

Arm 1 (Verum group): a treatment arm where the participant will receive homeopathic consultation plus a homeopathic remedy Arm 2 (Placebo group): a treatment arm where the participant will receive homeopathic consultation plus a placebo remedy Arm 3 (Usual care group): participants will continue with usual care and will not receive homeopathic treatment as part of the study.

Participants enrolled in this study, regardless of which study Arm they are in, may continue with all conventional medications or any other aspect of their current standard of care they are taking as recommended by their usual physician (so long as they are on a stable dose of the conventional ADHD medication for at least 6 weeks prior to beginning the trial). They may also continue to attend regularly scheduled visits with their own health care practitioner(s).

Participants may also start, stop or change the dose of any therapy (including conventional medications) during the study and are asked to report the change to the study team. Thus, the placebo group participants are not different than other participants, except that they will have a homeopathic consultation and a placebo remedy. The use of placebo is specific to homeopathic treatment, to allow for double-blinding, which is recognized to reduce study bias.

Prior to enrolling in the study, those considering participation will undergo a full assessment by a psychiatrist with a specialty in child and youth mental health. This assessment confirms the diagnosis and screens for inclusion/exclusion study criteria. At the same time, the psychiatrist recommends evidence-based therapies to clients including conventional medication. The psychiatrist does not directly treat the client. If medication is recommended and the clients wish to pursue it with their regular physician, they would still be able to enroll in the study if they wanted to, after six weeks of reaching a stable dose.

This study will help our understanding of the treatment process and whether different elements of the intervention have greater or lesser effects.

This study is a follow-up to an open label pilot study of the homeopathic treatment of ADHD using the same study team. Sample size was calculated based on the results of that study.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of attention deficit hyperactivity disorder (and any of the subtypes of the diagnosis) confirmed by study psychiatrist
* have a minimum baseline score on the Connors 3 scale that is 1.5 standard deviations above the population norm based in the age and sex of the participant as was reported to be most commonly used in ADHD treatment trials
* are between 6 and 16 years of age
* are able to ingest medications in liquid or in lactose/sucrose granule form;
* if currently taking stimulant therapy for ADHD, are on a stable dose for a minimum of 6 weeks prior to beginning the study
* have an estimated I.Q. within the normal range
* have parents/guardians who are able to read and write in English

Exclusion Criteria:

* a diagnosis with an additional mental health disorder including, but not limited to, the following: Conduct Disorder, Autism Spectrum Disorder, Bipolar Disorder, and Major Depressive Disorder
* any significant suicidality
* an addiction to any substance
* taking any other prescription medication aside from a stable dose of ADHD medication
* a history of head injury (with sequelae), seizures, or organ system damage
* pregnant or lactating

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Conners 3 Global Index - Parent | Baseline and weeks 8, 20, 28

SECONDARY OUTCOMES:
Change from baseline in Conners ADHD Index Probability score | Baseline and weeks 8, 20, 28
Change from baseline in Conners Content Scale for Inattention and Hyperactivity/Impulsivity | Baseline and weeks 8, 20, 28
Change from baseline in Conners DSM-IV-TR Symptom Scale for the ADHD Inattentive and ADHD Hyperactive-Impulsive subtypes | Baseline and weeks 8, 20, 28
Clinical Global Impression-Improvement scale | Week 28
Change from baseline in the Pediatric Quality of Life Inventory | Baseline and weeks 8, 20, 28
Change from baseline in Consultation and Relational Empathy measure | Baseline and weeks 8, 20, 28
Change from baseline in RTI Provider Support Measure | Baseline and weeks 8, 20, 28
Change from baseline in the Resiliency Scales for Children & Adolescents - Mastery sub-scale | Baseline and weeks 8, 20, 28
Change from baseline in Coping Efficacy Scale | Baseline and weeks 8, 20, 28
Change from baseline in Control Beliefs Inventory - Mastery sub-scale | Baseline and weeks 8, 20, 28

CONTACTS AND LOCATIONS:
Overall Officials: Heather Boon, PhD, Principal Investigator — University of Toronto
Locations (1):
- Riverdale Homeopathic Clinic, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Brule D, Landau-Halpern B, Nastase V, Zemans M, Mitsakakis N, Boon H. A Randomized Three-Arm Double-Blind Placebo-Controlled Study of Homeopathic Treatment of Children and Youth with Attention-Deficit/Hyperactivity Disorder. J Integr Complement Med. 2024 Mar;30(3):279-287. doi: 10.1089/jicm.2023.0043. Epub 2023 Sep 6. PMID 37672605